CLINICAL TRIAL: NCT00663559
Title: Study Phase II to Determinate the Efficacy of Sunitinib in Patients With Renal Cells Carcinoma Metastasic or Locally Avanced in Patients Not Candidates to Curative Previous Nefrectomy
Brief Title: Sunitinib in Patients With Renal Cells Carcinoma Metastasic or Locally Avanced in Patients Not Candidates to Curative Previous Nefrectomy
Acronym: SOGUG/0107
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG/0107
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2007-11

CONDITIONS: Carcinoma Renal Cells
Keywords: renal; Sunitinib; Unresectable and/or metastatic renal cell cancer
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): This study has only one arm with Sunitinib
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50mg oral in the morning during 4 weeks with 2 weeks of break.
  Other Names: Sutent

SUMMARY:
The purpose of this trial is to determinate the efficacy of Sunitinib in patients with renal cells carcinoma metastasic or locally avanced in patints not candidates to inicial curative nefrectomy.

DETAILED DESCRIPTION:
Study phase II in with one arm in patients with renal cells carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give their written informed consent before any procedure related to the study is performed.
* Patients with renal clear cell carcinoma metastatic or locally advanced, histologically or cytologically documented.The patients with metastasic disease must be not condidated to curative nefrectomy as investigator criteria.
* Assessable or measurable disease according to RECIST criteria. The lesions previosly radiated is not considered as target.
* Ages equal or superior to 18 years old.
* ECOG ≤ 1
* Patients with a life expectancy superior to 12 weeks.
* Patients with adequate organic function, according to the following criteria:

  1. . Medular reserve: Neutrophils absolute count≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Haemoglobin ≥ 9g/dl
  2. . Hepatic function: Total bilirubin < 1.5 times the superior limit of normality ALT and AST < 2.5 times the superior limit of normality (< 5 times the superior limit of normality in case of liver failure due to cancer)
  3. . Seric Albumin ≥ 1.5 times the superior limit of normality
  4. . Renal Function: Cleary creatinine > 30ml/min
  5. . FEVI > LIN according to ECO or MUGA
* Patients who are capable of accomplishing the study's requirements and without any impediments to follow the instructions while on study

Exclusion Criteria:

* Pregnant or breastfeeding women. Women of fertile age must have a negative result in the pregnancy test performed 7 days before the beginning of the administration of the study medication. Both men and women included in the study must use an adequate contraceptive method.
* Patients that have received sistemic treatment previous to metastasic disease.
* Previous nefrectomy.
* Mayor Surgery, radiotherapy or sistemic therapy received in the last 3 weeks previous to the inclusion of the patient in the study, except paliative radiotherapy upper no target lesions.
* Radiotherapy upper > 25% bone marrow.
* Patients that are participating in any clinical trial.
* Patients with a primary cancer diagnosis in thast 3 years, except superficial basaliomas, superficial escamous carcinoma or in situ cervix carcinoma with aducuate treatment.
* Following events in the last 12 months previous to begin the treatment: myocardial infarction, unstable o severe angina, coronary/periferic place of arterial by-pass, congestive cardiac insufficiency, brain-vascular accident included transitory ischemia or lung embolism.
* Arterial uncontrolled hypertension nor controlated with drugs ( >150/100 mmHg despite adequate medical treatment).
* Cardiac arrhythmia with grade NCI CTCAE ≥2, auricular fibrillation all grade and/or QTc interval> 450mseg in men and > 470 mseg in women.
* Actually treatment with therapeutic dose with acenocumarol (except low dose for deep venous thrombosis).
* Patients that present previously known positive serology for HIV.
* Abuse of substances, clinical conditions, psychological or social, that may interfere with the patient's participation in the study or with the evaluation of the study's results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 12 weeks

SECONDARY OUTCOMES:
Global survival | At last contact date or death date
Response global | Every 12 weeks
Duration of response | Every 12 weeks
Security and tolerability of Sunitinib | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Luís González Larriba, MD, Study Chair — SOGUG
Locations (7):
- Spain (7):
  - Hospital CLINIC, Barcelona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital de Jaén, Jaén, Jaén
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital lozano Blesa, Zaragoza, Zaragoza